CLINICAL TRIAL: NCT00366158
Title: EVITA: Evaluation of VIP Feature in Pacemaker Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Christophe Bailleul, St. Jude Medical
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR06001LV
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmia
Keywords: Patients with intact AV conduction
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ventricular Instrinsic Preference (VIP) turned ON
  Interventions: Device: Device: St. Jude Medical Victory dual-chamber pacemaker; Device: Ventricular Intrinsic Preference
- 2 (Active Comparator): Ventricular Instrinsic Preference (VIP) turned OFF
  Interventions: Device: Device: St. Jude Medical Victory dual-chamber pacemaker; Device: Ventricular Intrinsic Preference

INTERVENTIONS:
Device: Device: St. Jude Medical Victory dual-chamber pacemaker — Pacemaker implant
Device: Ventricular Intrinsic Preference — Programming of pacemaker

SUMMARY:
The primary efficacy objective of this clinical investigation is to demonstrate that the Ventricular Intrinsic Preference (VIP™) feature allows to reduce the medium- and long-term incidence of unnecessary ventricular pacing in patients with intact AV conduction.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an indication for implantation of a dual-chamber pacemaker;
* Patient is implanted or scheduled to be implanted with a St Jude Medical Victory pacemaker, or newer device with the same study relevant feature.

Exclusion Criteria:

* Patient has persistent or permanent AF/AFl;
* Patient has permanent AV Block;
* Patient has a pacemaker replacement;
* Patient is in NYHA class IV;
* Patient is unable to attend the follow-up visits;
* Patient is pregnant;
* Patient is less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Percentage of ventricular pacing | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bauer, MD, Study Chair — Universitätskliniken Heidelberg, Heidelberg, 69115, Germany; Charles Kennergren, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Universitätskliniken Heidelberg, Heidelberg, Germany
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Bauer A, Vermeulen J, Toivonen L, Voitk J, Barr C, Peytchev P. Minimizing right ventricular pacing in pacemaker patients with intact and compromised atrioventricular conduction : Results from the EVITA Trial. Herzschrittmacherther Elektrophysiol. 2015 Dec;26(4):359-66. doi: 10.1007/s00399-015-0394-2. Epub 2015 Aug 28. PMID 26315154